CLINICAL TRIAL: NCT06562946
Title: An Open-Label, Parallel-Group, Single-Dose Study to Assess the Pharmacokinetics of Pimicotinib in Subjects With Mild and Moderate Hepatic Impairment Relative to Subjects With Normal Hepatic Function
Brief Title: The Study to Assess the Pharmacokinetics of Pimicotinib in Subjects With Mild and Moderate Hepatic Impairment Relative to Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ABSK021-106
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The mild (Child-Pugh score 5 to 6) hepatic impairment. (Experimental): Subjects will enter the study site on Day -1 and will remain there until after the collection of the 48 h PK samples on Day 3. On Day 1 all participants will receive a single 25 mg oral dose of pimicotinib under fasting conditions, followed by extensive blood collection and urine sample collection for measurement of pimicotinib and its metabolites.
  Interventions: Drug: Pimicotinib
- The moderate (Child-Pugh score 7 to 9) hepatic impairment. (Experimental): Subjects will enter the study site on Day -1 and will remain there until after the collection of the 48 h PK samples on Day 3. On Day 1 all participants will receive a single 25 mg oral dose of pimicotinib under fasting conditions, followed by extensive blood collection and urine sample collection for measurement of pimicotinib and its metabolites.
  Interventions: Drug: Pimicotinib
- The healthy subjects. (Experimental): Subjects will enter the study site on Day -1 and will remain there until after the collection of the 48 h PK samples on Day 3. On Day 1 all participants will receive a single 25 mg oral dose of pimicotinib under fasting conditions, followed by extensive blood collection and urine sample collection for measurement of pimicotinib and its metabolites.
  Interventions: Drug: Pimicotinib

INTERVENTIONS:
Drug: Pimicotinib — Pimicotinib is supplied as capsules for oral use with a strength of 25 mg/capsule.

SUMMARY:
This is a phase 1, open-label, parallel-group, single-center study to evaluate the pharmacokinetics and safety of a single 25 mg oral dose of pimicotinib in subjects with mild and moderate hepatic impairment and in control subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should understand the study procedures and sign the informed consent form prior to Screening.
2. Subjects must be 18 to 70 years of age inclusive, at the time of signing the informed consent.
3. Weight ≥ 50 kg for males and ≥ 45 kg for females, with a body mass index (BMI) between 18 and 32 (inclusive), BMI = weight (kg)/height (m)2.
4. Serum creatinine (Cr) ≤ 1.5 × ULN, or Creatinine clearance (Crcl) ≥ 60 mL/min (Cockcroft-Gault formula).

Exclusion Criteria:

1. Known allergy or hypersensitivity to any components of the investigational drug product;
2. Has a history of cancer in five years (malignancy), exceptions include cured basal cell carcinoma of skin, squamous cell carcinoma of skin, and other carcinomas in situ;
3. Has factors that significantly affect the absorption of oral drug, such as inability to take oral medication or significant nausea and vomiting, malabsorption, external bile duct drainage, massive small bowel resection, etc.
4. Has a history of portosystemic shunt.
5. Participation in any clinical study of an investigational drug/device within 3 months of the drug prior to Day -1;
6. Received live vaccines or live-attenuated virus vaccine within 3 months prior to screening, or plan to get vaccinated during the study;
7. Previously participated in this study or any other study related to pimicotinib and received pimicotinib;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Conduct testing within 2 month after all subjects collect all samples at all time points required by the protocol
  To evaluate the pharmacokinetics (PK) of pimicotinib and its two identified metabolites, M281 and M436-2, following a single oral dose of pimicotinib capsules in adult subjects with mild and moderate hepatic impairment compared to healthy control subjects.
AUClast | Conduct testing within 2 month after all subjects collect all samples at all time points required by the protocol
  To evaluate the pharmacokinetics (PK) of pimicotinib and its two identified metabolites, M281 and M436-2, following a single oral dose of pimicotinib capsules in adult subjects with mild and moderate hepatic impairment compared to healthy control subjects.
AUC 0-∞ | Conduct testing within 2 month after all subjects collect all samples at all time points required by the protocol
  To evaluate the pharmacokinetics (PK) of pimicotinib and its two identified metabolites, M281 and M436-2, following a single oral dose of pimicotinib capsules in adult subjects with mild and moderate hepatic impairment compared to healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yanan Wang, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No